CLINICAL TRIAL: NCT04140890
Title: Supporting Habit Formation to Attenuate Prefrailty in Elders: a Pilot Study
Brief Title: Supporting Habit Formation to Attenuate Prefrailty in Elders: Pilot Study
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Heather Fritz, Assistant professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 065319B3E
Record Dates: First submitted 2019-10-21; First posted 2019-10-28 (Actual); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Frailty
Keywords: prefrail; habit; exercise; diet
MeSH Terms: conditions — Frailty; Habits; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The treatment group will receive healthy habit intervention, and the control group will receive attention control.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants in the treatment group will be asked to meet with an occupational therapist in their home weekly over 12 weeks. Each session takes an hour. In the first session, the occupational therapist will introduce the program. In session 2, the therapist will discuss pain and pain management with the participant. In session 3-12, the therapist will help the participant to develop physical activity and healthy eating habits. In each session the participant will pick two healthy behaviors to turn them into a habit. The therapist will give the participant a workbook and teach the participant to track his/her progress. The focus of session 3-5 will be physical activity, and session 6-11 will be healthy eating. In the last session (session 12), the therapist will wrap up the program and help the participant to develop a maintenance plan.
  Interventions: Behavioral: Habit Formation
- Control (Placebo Comparator): Participants in the control group will receive newsletters focused on general healthy aging topics over 12 weeks. With the exception of two, 1-page handouts covering PA and dietary recommendations, the weekly content will not overlap with the treatment content. Within 4 days of mailing the newsletter, a trained research assistant (RA) will call the participant, verify receipt of the newsletter, and ask them if they have any questions about the materials. The phone call will last ~15 minutes. Control condition participants receive no further intervention.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Habit Formation — Treatment sessions consist of 12 weekly health coaching sessions at participants' home. During the intervention period, an occupational therapist will help the participant to commit to developing new simple habits (dietary habits or physical activity habits) in each 60-minute session.
  Arms: Treatment
Behavioral: Education — In the education group, participants will receive newsletters containing general healthy aging materials over 12 weeks. A trained research assistant will call participants to verify receipt of the newsletter, and answer their questions about the materials. Each phone call will last ~15 minutes.
  Arms: Control

SUMMARY:
The Supporting Habit Formation to Attenuate Prefrailty in Elders (SHAPE) Pilot Study is a randomized control study. The main objective of this pilot study is to determine the feasibility of using Habit Formation (HF) treatment to increase Physical Activity (PA) (reduction in daily in hours of sedentary time), and dietary among prefrail African Americans. We hypothesize: (1)The SHAPE study will demonstrate good feasibility with a high recruitment rate and successful administration all of the measures among the target population; (2) Treatment group participants will demonstrate greater increases in primary outcomes (physical activity level and dietary quality) and secondary outcomes (quality of life, depressive symptoms, prefrailty reduction, lower extremity strength and balance, physical activity level, waist circumference, and weight at intervention completion.

DETAILED DESCRIPTION:
Frailty signifies a decline in physical, cognitive and/or psychosocial reserve that reduces an older adult's ability to respond to or recover from stressors (e.g., acute illness) and contributes to early morbidity and mortality. Nearly half of all older adults are prefrail, and prefrailty status increases the risk of becoming frail. Frailty is more prevalent among African Americans and occurs earlier in life when compared to European Americans. Older African Americans in the US, face significant challenges in adhering to frailty reduction treatment such as increasing physical activity (PA) and adopt a healthy diet. Those challenges include poverty, accelerated aging, higher levels of activities of daily living disability, and less access to safe opportunities for PA or healthy food. The situation is even worse for urban-dwelling older African Americans, who often reside in neighborhoods replete with physical and social stressors (e.g., derelict infrastructure or crime) that intersect with the vulnerabilities of aging, to further complicate their efforts to engage in frailty protective behaviors. Despite this, frailty interventions overwhelmingly exclude African Americans, thereby limiting generalizability to this high-risk group.

Therefore, the rationale of this study is to test the feasibility of a novel habit formation (HF) intervention to facilitate frailty protective behaviors in prefrail African Americans ages 55 and older in a randomized control trial study. The HF intervention targets two main health behaviors: decrease sedentary time (ST) and improve dietary quality. The intervention consists of 12 treatment sessions over 12 weeks. In each session, an occupational therapist will deliver educational content, and use HF techniques and behavioral skills to facilitate frailty protective behaviors. Forty-eight prefrail African American adults will be randomized to the treatment or control group. The baseline evaluation will be conducted before randomization and the follow-up evaluation after the last treatment session. For the treatment group participants, we will further evaluation occupational activity performance/satisfaction and habit formation strength within treatment sessions.

The main goal of this study is to determine the feasibility of HF intervention among prefrail African American adults. The main hypothesis is: the SHAPE study will demonstrate good feasibility with (1) high recruitment rate (recruit 48 participants over 6 months), (2) treatment group participants will show preliminary efficacy in primary outcomes such as reducing sedentary time (measured by the ActivPal device) and increasing dietary quality score (measured by Healthy Eating Index [HEI]) at intervention completion compared to controls. The secondary hypothesis is: treatment group participants will demonstrate preliminary efficacy in secondary outcomes such as increased quality of life (measured by the Cardiovascular Health Study frailty criteria), reduced depressive symptoms (Geriatric Depression Short form), prefrailty reduction (The Fried's Frailty Criteria Index), increased lower extremity strength and balance (Short Physical Performance Battery), increased physical activity level (The Community Healthy Activities Model Program for Seniors), reduced waist circumference and weight at intervention completion compare to controls.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Community-dwelling
* Prefrail (evaluated by the Frailty scale)
* Self-identify as African Americans.

Exclusion Criteria:

* Diagnosed psychiatric disorders,
* Moderate or severe cognitive impairment (using the Six Item Cognitive Impairment Test and operationalized as a score of ≥ 10),
* Using prescription drugs that could affect cognition and functioning (e.g., neuroleptics), - - Individuals with typical daily pain ratings of ≥ 7/10 on a 10 point Likert scale of pain
* Planing to change residences during the study period
* Relying on a wheelchair for home or community mobility
* Actively receiving home care services, occupational, or physical therapy
* On dialysis or who have an end of stage disease (e.g., stage IV heart failure)
* Enrolling in a health promotion program focused on physical activity and diet
* Have a baseline healthy eating index score of ≥ 85/100 as their diet would already be very close to ideal (average score for U.S. population = 59)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Fritz, PhD, Principal Investigator — Wayne State University
Locations (1):
- Eugene Applebaum College of Pharmacy and Health Sciences, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from September 2019 to March 2020 in metropolitan Detroit, Michigan.
Pre-assignment Details: Drop out due to unable to comply to study procedure (n=4) Disenroll due to COVID-19 outbreak (n=5)
Period: Overall Study
Arm/Group | Treatment | Control
Started | 9 | 12
Completed | 9 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (12.4) | 74.6 (8.1) | 73.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completed the Study
Description: The number of participants completed the intervention and post-test.
Time Frame: baseline to 6 months
Population: Contacted 30 participants before the intervention started.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 15 | 15
Participants | 9 | 11

2. Primary Outcome: Seven-days Average Sedentary Time (Minutes/Day)
Description: A physical activity tracking system activPAL™. The ActivPal sensor will be attached to participants' thigh for 7 consecutive days.
Time Frame: baseline to 14 weeks
Population: One treatment group participant was excluded because the participant did not complete the full assessment at post-test.
Measure: Mean (Standard Deviation); unit: min/day
Arm/Group | Treatment | Control
Number analyzed (Participants) | 8 | 11
min/day
  Pre-test | 551.9 (128.1) | 555.5 (166.4)
  Post-test | 565 (129.7) | 582.3 (191)

3. Primary Outcome: Healthy Eating Index Score
Description: ASA 24 is a web-based tool for participants to recall their diet on a daily basis. The HEI score is calculated by a standard SAS code provided by ASA 24 website to evaluated the content of participants' dietary recalls. Scores range from 1-100 with higher scores indicating better quality diet.
Time Frame: Baseline to 14th week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 9 | 11
score on a scale
  Healthy eating index score at pre-test | 44.4 (17.4) | 46.7 (11.9)
  Healthy eating index score at post-test | 46.9 (14.3) | 46.9 (7.5)

4. Secondary Outcome: The The World Health Organization Quality of Life- BREF
Description: The World Health Organization Quality of Life- BREF (WHOQOL-BREF) is a 26 item questionnaire, which measures the four broad domains of quality of life(QOL): physical health, psychological health, social relationships, and environment. Items are rated on a 5-point Likert scale (low score of 1 to a high score of 5) to determine a raw item score. Subsequently, the mean score for each domain is calculated, resulting in a mean score per domain that is between 4 and 20. To compare the results with other studies, the mean scores per domain is then converted into transformed scores based on the WHOQOL-BREF scoring manual. The transformed scores per domain range from 0 to 100, where a higher score indicates better QOL.
Time Frame: Baseline to 14th week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 9 | 11
score on a scale
  Physical at pre-test | 78.1 (18.5) | 72.7 (12.5)
  Physical at post-test | 78.6 (16.6) | 73.1 (15.8)
  Psychological at pre-test | 72.2 (14.9) | 83.3 (8.9)
  Psychological at post-test | 74.1 (20) | 81.1 (8.2)
  Social Relationship at pre-test | 63.9 (15.6) | 82.6 (8.7)
  Social Relationship at post-test | 63.9 (22.1) | 73.5 (14.4)
  Environment at pre-test | 73.6 (19.1) | 79.8 (11.6)
  Environment at post-test | 72.6 (23.8) | 83 (9.9)

5. Secondary Outcome: Geriatric Depression Short Form (GDS)
Description: The Geriatric Depression Short form (GDS) is a 15-item measure in which participants self-report depressive feelings (scoring range from 0-15). A higher score indicates more depressive symptoms.
Time Frame: Baseline to 14th week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 9 | 11
score on a scale
  Pre-test | 2.3 (2.5) | 1.3 (0.8)
  Post-test | 3.9 (4.2) | 1.6 (1.4)

6. Secondary Outcome: The Fried's Frailty Criteria Index
Description: The Fried's Frailty index is a 5-item measure indicating the number of frailty symptoms (scale range from 0-5). A higher score indicates more frailty symptoms (worse outcomes).
Time Frame: Baseline to 14th week
Population: One treatment group participant was excluded because the participant did not complete the full assessment at post-test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 8 | 11
units on a scale
  Pre-test | 1.9 (1.5) | 0.9 (1)
  Post-test | 1.6 (1.4) | 0.9 (0.7)

7. Secondary Outcome: Short Physical Performance Battery (SPPB)
Description: The Short Physical Performance Battery-Balance Test (SPPB) assess balance and mobility with three subtests (score range: 0 to 4): standing balance, three-meter gait speed, and five repetitions of sit-to-stand motion. Total score are sums of subtest scores ranging from 0 (worst performance) to 12 (best performance).
Time Frame: Baseline to 14th week
Population: One treatment group participant was excluded because the participant did not complete the full assessment at post-test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 8 | 11
score on a scale
  Pre-test | 6.8 (2.8) | 7.1 (2.4)
  Post-test | 7.6 (2.2) | 7.3 (2.5)

8. Secondary Outcome: The Community Healthy Activities Model Program for Seniors (CHAMPS)
Description: The CHAMPS is 41-item, self-administered instrument assessing physical activity patterns among older adults. Each item asks for the frequency and duration of an activity that older adults do in the past week. Energy expenditure (Kcal/week) of physical activities is calculated from the items.
Time Frame: Baseline to 14th week
Measure: Mean (Standard Deviation); unit: kcal/week
Arm/Group | Treatment | Control
Number analyzed (Participants) | 9 | 11
kcal/week
  Pre-test | 1915.6 (2063.5) | 2014.4 (1912.3)
  Post-test | 2694.5 (1761.1) | 1838.1 (781.3)

9. Secondary Outcome: Waist Circumference
Description: Waist circumference in inches is measured by the Gulick II tape measure.
Time Frame: Baseline to14th weeks
Population: One treatment group participant was excluded because the participant did not complete the full assessment at post-test.
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | Treatment | Control
Number analyzed (Participants) | 8 | 11
Inches
  Pre-test | 40.8 (3.2) | 39.7 (4.8)
  Post-test | 40.1 (4.5) | 40 (4.4)

10. Secondary Outcome: Weight
Description: Weight (pounds) is measured by medical weight scales.
Time Frame: Baseline to 14 weeks
Population: One treatment group participant was excluded because the participant did not complete the full assessment at post-test.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Treatment | Control
Number analyzed (Participants) | 8 | 11
pounds
  Pre-test | 172 (34.3) | 177.8 (37.7)
  Post-test | 172.5 (32.3) | 179.5 (35.1)

11. Other Pre Specified Outcome: The Canadian Occupational Performance Measure (Treatment Group Only) (COPM) for Treatment Group Only
Description: The COPM is self-perception of occupational performance in the areas of self-care, productivity and leisure. The COPM is administered using a semi-structured interview in which the client identifies significant issues in daily activities which are causing difficulty. The importance of each activity, as perceived by the client, is first rated on a 10-point scale ranging from 1 (not important at all) to 10 (extremely important). In the next step the client selects the five most important activities, which are then rated on a 10-point scale for performance, ranging from 1 (not at all able) to 10 (able to perform extremely well), and for satisfaction, ranging from 1 (not at all satisfied) to 10 (extremely satisfied). Increased performance/satisfaction score from follow-up to baseline represents improved performance/satisfaction.
Time Frame: Pre-test to week 13
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Treatment: Participants in the treatment group will be asked to meet with an occupational therapist in their home weekly over 12 weeks.
Arm/Group | Treatment
Number analyzed (Participants) | 9
score on a scale
  Performance at pre-test | 4.6 (2.0)
  Performance at post-test | 5.3 (2.3)
  Satisfaction at pre-test | 3.6 (2.4)
  Satisfaction at post-test | 5.7 (2.8)

12. Other Pre Specified Outcome: The Modified Self-reported Habit Index (Treatment Group Only)
Description: The modified self-reported habit index (SRHI) is a 4-item assessment that measures habit strength, frequency, relevance to self-identity, and automaticity. Items are self-rated with a seven-point Likert scale (1=strongly disagree, 7= strongly agree). The average score of the 4 items range from 1 to 7 indicates habit formation, where higher scores indicate stronger the habit is. During 9 treatment sessions (the 3,4,5,6,7,8,9,10,11 treatment sessions), 2-4 habits regarding physical activity and diet will be assessed individually with the modified SRHI. Post-test of each habit will be assessed again after 2 weeks. We calculated the average score of the index of each habit.
Time Frame: baseline to two weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 9
score on a scale
  Pre-test | 1.89 (0.87)
  Post-test | 4.69 (1.24)

ADVERSE EVENTS:
Time Frame: The adverse event of each participant was monitored from baseline to 14 weeks, starting from baseline evaluation.
Description: The risk of this study is minimal to the participants.
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT04140890/Prot_SAP_000.pdf